CLINICAL TRIAL: NCT02481011
Title: Risk of Intracranial Hemorrhage in Users of Oral Antithrombotic Drugs: a Nationwide Study
Brief Title: Risk of Intracranial Hemorrhage in Users of Oral Antithrombotic Drugs
Acronym: RICH
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/7958
Record Dates: First submitted 2015-06-22; First posted 2015-06-25 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Intracranial Hemorrhages; Stroke
Keywords: Fibrinolytic agents; Adverse effects; Registries; Incidence; Risk assessment
MeSH Terms: conditions — Intracranial Hemorrhages; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- users: patients on antithrombotic drugs admitted to a Norwegian hospital for intracranial hemorrhage (ICH)
  Interventions: Drug: antithrombotic drugs
- non-users: patients not on antithrombotic drugs admitted to a Norwegian hospital for intracranial hemorrhage (ICH)

INTERVENTIONS:
Drug: antithrombotic drugs
  Groups: users

SUMMARY:
The true incidence and risks of intracranial hemorrhage (ICH) in patients on various antithrombotic treatments remain unknown. Here a nationwide study is conducted to investigate the risk for and incidence rates of ICH in users and non-users of various oral antithrombotic drugs in Norway between 2008 through 2014.

Hopefully, this study will contribute to a more responsible prescription pattern of antithrombotic medications.

DETAILED DESCRIPTION:
The most serious adverse effect of antithrombotic therapy is bleeding. Combinations of antithrombotic agents are now frequently used (e.g. after use of drug eluting stents or after ischemic stroke), and this may lead to an increased frequency of significant bleeding complications. Among hemorrhagic complications of antithrombotic drugs, intracranial hemorrhage (ICH) may have particularly devastating consequences with high morbidity, disability and even mortality rates. Intracerebral hemorrhage (hemorrhagic stroke) is generally associated with a higher risk for death and incurs greater loss of health over a lifetime than ischemic stroke.

This makes antithrombotic therapy a double-edged sword. Although a certain risk for bleeding may be acceptable in the context of even greater protection against ischemic events, it is important to quantify the magnitude of bleeding risk. So far the efficacy and safety profile of antithrombotic agents are generally assessed in randomized controlled trials (RCT). However, extrapolating the results from randomized clinical trials to the general patient population in this context is challenging. Patients who participate in clinical trials are frequently highly selected and therefore somewhat unrepresentative. In addition, their numbers are limited and the treatment period is often much shorter than in routine management of a chronic disease or condition. Finally, patients in clinical trials are often monitored more closely than in routine practice.

The incidence of intracranial hemorrhage due to antithrombotic therapy could theoretically be monitored by post-marketing surveillance by including spontaneously reported events. Unfortunately, it seems this does not provide more reliable estimates. A recent study from Finland has shown that bleeding complications due to oral anticoagulation with Warfarin are underreported in daily clinical practice. Further, it has been shown that reporting rates of side effects following medical therapy tend to decrease over time indicating that it is more likely that adverse events to a newer drug are reported than to a drug that has been available for many years. This is why population-based large-scale pharmaco-epidemiological studies are needed, in which cohorts of patients exposed to antithrombotic medications are monitored to determine a valid and reliable risk of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* hospitalization due to intracranial hemorrhage (ICH)
* residential address in Norway

Exclusion Criteria:

* Traumatic (high-energy) intracranial injury
* Parenteral antithrombotic treatment
* ICH related to tumor or vascular malformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with intracranial hemorrhage admitted to hospitals in Norway 2008-2014
Sampling Method: Non-Probability Sample
Enrollment: 22111 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
incidence rate of intracranial hemorrhage (ICH) requiring hospitalization | 6 years
  We will determine the incidence rates of ICH in users and non-users of oral antithrombotic treatment by linking data from Norwegian Patient Register (NPR) and the Norwegian prescription database.

SECONDARY OUTCOMES:
overall survival following ICH | 6 years
  comparison of users and non-users of oral antithrombotic drugs
proportion of ICH patients undergoing neurosurgical procedures | 6 years
  comparison of users and non-users of oral antithrombotic drugs

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Gulati, md phd, Study Director — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Background] Gulati S, Solheim O, Carlsen SM, Oie LR, Jensberg H, Gulati AM, Giannadakis C, Jakola AS, Salvesen O. Risk of intracranial hemorrhage in users of oral antithrombotic drugs: Study protocol for a nationwide study. F1000Res. 2015 Dec 30;4:1519. doi: 10.12688/f1000research.7633.1. eCollection 2015. PMID 26918124
- [Result] Gulati S, Solheim O, Carlsen SM, Oie LR, Jensberg H, Gulati AM, Madsbu MA, Giannadakis C, Jakola AS, Salvesen O. Risk of intracranial hemorrhage (RICH) in users of oral antithrombotic drugs: Nationwide pharmacoepidemiological study. PLoS One. 2018 Aug 23;13(8):e0202575. doi: 10.1371/journal.pone.0202575. eCollection 2018. PMID 30138389